CLINICAL TRIAL: NCT02193386
Title: Evidence-based Practice and Its Effectiveness in Physical Therapy Treatment of Children With Bilateral Spastic Cerebral Palsy.
Brief Title: Evidence-based Physical Therapy in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: S51880; ML5982 (Registry Identifier: UZ Leuven)
Record Dates: First submitted 2014-07-10; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2010-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Physical Therapy; gait analysis; gross motor function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): No intervention, no follow-up, only registration of usual therapy
  Interventions: Other: No intervention, no follow-up, only registration
- Intervention period (Experimental): Predefined, evidence-based program and support
  Interventions: Other: Intervention period

INTERVENTIONS:
Other: No intervention, no follow-up, only registration — Usual Care
  Arms: Usual Care
Other: Intervention period — Predefined intervention program
  Arms: Intervention period

SUMMARY:
The study aims to evaluate evidence-based practice behavior in usual care physical therapy in Flanders. Secondly, it aims to compare the effectiveness of a predefined physical therapy program based on evidence-based guidelines to the effects of a period of usual care. It is hypothesized that supporting therapists by providing a predefined evidence-based intervention program, will result in an improved treatment outcome compared to the usual care physical therapy.

DETAILED DESCRIPTION:
Participants A convenience sample of 16 children will be recruited at the Cerebral Reference Centre of the University Hospital Pellenberg. Children will be included when they are diagnosed with bilateral spastic CP, aged between 4 and 9 years and a Gross Motor Function level between I and III. Children are excluded when they received Botulinum Toxin A injections within the past six months, orthopedic surgery in the past or had severe associated problems that limited participation to therapy (blindness, deafness, severe cognitive limitations or autism).

Design All children will start the study with a registration period. During this period, the children's usual physical therapy (UC) will be registered using a diary. Immediately following the UC period, children will be enrolled into a predefined intervention program (IP).

Both the period of UC and IP will have a duration of 10 weeks. Before and after both periods, children will be evaluated using the Gross Motor Function Measurement (GMFM-88) and three-dimensional gait analysis (3DGA).

Therapy interventions During the period of UC, no specific intervention will be provided. Children will receive the frequency, intensity and contents of therapy as they usually receive by their own private physical therapist. A diary will be provided to the child's physical therapist. The diary contains session forms, designed for the therapist to carefully register the contents of therapy after each session.

In the session forms, the therapist will note down how much time of the therapy session will target problems at the different levels of the ICF. At the level of body structure and function, the time spent on muscle length and muscle strength will be registered. For muscle length, the therapists are asked to report the targeted muscles, the number of repetitions, the duration of stretch and treatment modality (activo, activopassivo or passivo). About muscle strength, therapists will note the specific muscle that was trained, the intensity (number of repetitions and resistance) and whether the exercise was performed as analytical (single-joint) or functional (multiple-joint) muscle work. Concerning activity level, the specific functional activity that was practiced and the averaged position in which this was performed, will be registered. Finally, the therapist will be asked to report whether any problems at participation level are specifically addressed.

During the period of UC, the therapist will not be contacted and no instructions or advice will be provided regarding physical therapy treatment of the child.

Intervention period

Immediately following the UC period, children were enrolled into a predefined intervention program (IP), designed by the first and third author of the study. The programs will be executed by the child's personal physical therapist, who will agree to precisely follow the prescribed program. Similar as for the UC program, the children will receive the frequency of therapy as they usually receive by their own private physical therapist. Two different types of programs were designed. Ten children received an individually defined, targeted program tailored to the individual needs of the child and six children received a general program based on general age-appropriate treatment aims for children with bilateral spastic CP. For an extensive description of the differences and similarities between both types of intervention programs, the authors refer to our previous intervention studies. All intervention programs have two major common features. The first central and common aspect in the intervention programs was that basic principles regarding evidence-based training were respected. All programs consist of a predefined set of exercises to improve strength, selectivity and mobility and a set of functional exercises. Thereby, stretching is prescribed as three repetitions of 30 seconds and strength training was prescribed in series of three times 12 to 15 repetitions. Functional exercises are not restricted to a specific repetition number. As appropriate, all intervention programs will contain more than 50% of exercises at activity and participation level. The second major common feature in the intervention programs is the support and follow-up to the therapist. At the start of the intervention study, therapists will be visited and the prescribed program will be thoroughly explained. All exercises will be provided in a clear and structured way, with specific instructions regarding anatomical position, sets and repetitions. The specific exercises will be discussed and demonstrated if necessary. During the second or third week, the therapist will be contacted by phone or email to discuss the progress of the program and the possible needs to change and adjust exercises. Additionally, a follow-up visit will be organized around halfway through the program. During this visit, the program will again discussed and the therapist performed a regular therapy session using the program, in attendance of the first author of the study. Difficulties in performance were discussed and if necessary, some exercises were demonstrated. The opportunity for feedback on handling or position was thereby provided.

Due to these common aspects in our programs, and because previous data analysis revealed that the overall effects of both programs were not found to be significantly different, we can test our hypothesis regarding the influence of evidence-based support on the pooled data-set.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* Age 4- 9 y
* Gross Motor Function Classification I-III (ambulant)

Exclusion Criteria:

* Severe associated problems limiting participation to the programs
* Severe musculoskeletal limitations

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure - 88 | baseline, after 10 weeks of usual care and after 10 weeks of intervention

SECONDARY OUTCOMES:
Change in three-dimensional gait analysis | baseline, after 10 weeks of usual care and after 10 weeks intervention
  Gait Profile Score, Movement Assessment Profiles and time-and distance parameters

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven (Pellenberg) - Reference centre for children with Cerebral Palsy, Pellenberg, Flanders, Belgium